CLINICAL TRIAL: NCT05240768
Title: Clinical Outcomes of Patients With Deferred Revascularization Based on Fractional Flow Reserve (FFR) and Instantaneous Wave-free Ratio (iFR) Negative Coronary Artery Lesions in Pakistani Population
Brief Title: Clinical Outcomes of Patients With Deferred Revascularization Based on FFR and iFR Negative Coronary Artery Lesions.
Status: Completed | Type: Observational
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Jamshed Ali, Resident, Section of Cardiology, Department of Medicine, Aga Khan University Hospital, Pakistan
Other Study IDs: 2020-3681-10742
Record Dates: First submitted 2021-11-03; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Fractional flow reserve, instantaneous wave-free Ratio — Clinical outcomes observed for patients with moderate coronary lesions in whom coronary revascularization was deferred due to a negative physiologic study.

SUMMARY:
The objective is to assess long-term clinical outcomes of patients in whom intervention of coronary lesions was deferred due to negative fractional flow reserve (FFR) and negative Instantaneous wave-free ratio (iFR) in a real-world patient population and to identify factors associated with deferred target lesion failure.

DETAILED DESCRIPTION:
Fractional flow Reserve (FFR) evaluates functional significance of stenosis in intermediate coronary lesions. Instantaneous wave-free ratio (iFR) is considered noninferior to FFR and does not require adenosine administration.

This study was done to assess long-term clinical outcomes and factors associated with target vessel revascularization (TVR) in patients with deferred revascularization based on negative FFR and iFR.

Retrospective analysis of medical records of 345 patients with deferred revascularization at a tertiary care hospital , from January 2012 to January 2020 will be done.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had intermediate to severe coronary lesions on coronary angiogram.
* Patients who had negative FFR >0.80 or iFR >0.89 and did not undergo immediate or planned revascularization on basis of negative physiologic assessment.

Exclusion Criteria:

* Patients younger than 18 years of age or those having positive FFR/iFR values irrespective of revascularization status were excluded.
* Similarly, those who were lost to follow up and could not be traced via telephonic or were also excluded.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Mean age of study population was 62 ±11 years and majority (71%) of the population was male.76% (263) of the population was hypertensive, diabetes mellitus and dyslipidemia was present in 49%(169) and 53%(185) respectively. History of myocardial infarction (MI) was present in 12% (43) and one-fourth of population had history of revascularization, i.e PCI (19%) or coronary artery bypass grafting(CABG) 3%.
Sampling Method: Non-Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Cardiac death | 29 months
  Number of participants who died due to sudden cardiac arrest, sudden death due to acute MI and death due to heart failure or cardiogenic shock
Non-fatal myocardial infarction | 29 months
  Number of patients suffering from Myocardial infarction but did not die.
Target vessel revascularization. | 29 months
  Repeat PCI or bypass graft placement for a stenosis in another part of the vessel treated at the index PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan